CLINICAL TRIAL: NCT00347516
Title: Comparative Study of Three Intraocular Lens Power Calculation Formulae for Asian Eyes With Axial Lengths Less Than 22mm and Greater Than 25mm
Brief Title: Comparative Study of Three IOL Power Calculation Formulae for Asian Eyes Shorter Than 22mm or Longer Than 25mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Eye Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R430/25/2005
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Cataract
Keywords: IOL formula; High myopia; axial length
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Procedure: IOL calculation formula

SUMMARY:
Implantation of an intraocular lens is the gold standard in modern day cataract surgery.

The appropriate lens power needed to achieve the desired refractive outcome can be calculated with a whole variety of formulas.

To date, there has been no prospective study conducted to evaluate the accuracy of the IOL power calculation formulae commonly in use. It is well established that the frequently used IOL formulas do not show significant differences when used in eyes of average axial length (i.e. between 22mm and 25mm) and it is at the extremes of axial lengths where discrepancies arise. Our aim is to find the most appropriate formula(e) for these 'long' and 'short eyes' particularly in our population where there is a significant proportion of high myopes.

DETAILED DESCRIPTION:
Our primary objective is to compare three IOL power calculation formulae and determine the most appropriate formula for accurate prediction of postoperative refractive error in Asian eyes with axial length less than 22mm and greater than 25mm that are undergoing phacoemulsification cataract surgery.

This will be a randomized prospective study in patients with axial lengths less than 22mm and greater than 25mm undergoing phacoemulsification cataract surgery and IOL implantation. Each patient will be randomly assigned to have their IOL power calculated using one of three IOL power calculation formulae (SRK-T, Hoffer Q and Holladay 2). A randomization list will be used to decide the IOL formula allocation.

The primary outcome measure of this study is the mean absolute error (MAE) which is calculated by subtracting the intended formula-derived preoperative refractive error from the actual postoperative refractive error.

Based on the estimates from a previous study, it is postulated that the MAE for Hoffer Q, Holladay 2, and SRK-T are +0.36 D, +0.53 D & +0.74 D, respectively.

The interest here is pair-wise comparisons amongst SRK-T, Hoffer Q and Holladay 2. The sample size calculations for each pair-wise comparison is based on a SD of 0.57 D with a power of 80% and a 2-sided test of 5%. Using equal randomization, a total of 176 subjects would be sufficient to achieve statistical differences between Hoffer Q over the Holladay 2 & SRK-T and also the Holladay 2 over SRK-T (standardized effect difference of 30% between Hoffer Q & Holladay 2; 67% & 37% effect size for Hoffer Q vs SRK-T and Hollady 2 vs SRK-T, respectively).

Factoring in an attrition rate of 20%, a total sample size of 210 eyes will be recruited for the study.

Preoperatively, Snellen visual acuity will be assessed and all patients will undergo a non-cycloplegic autorefraction, keratometry measurement and axial length measurement with the Zeiss IOL Master (see below Visit 1). All patients will undergo phacoemulsification and 'in-the-bag' IOL implantation (Visit 2). Surgery will be performed through a 2.75mm temporal clear corneal incision and only the Alcon MA60BM or MA60MA 3-piece acrylic foldable IOL will be implanted. A standard postoperative topical antibiotic and anti-inflammatory regime consisting of tobramycin and beclomethasone will be administered (Visit 3-5).

Patients will be examined at the following intervals:

Screening Within 90 days prior to surgery Preoperative (Visit 1) Within 30 days prior to surgery Operative (Visit 2) Day of surgery Postoperative (Visit 3) 1 day after surgery Postoperative (Visit 4) 3-5 days after surgery Postoperative (Visit 5) 4-5 weeks after surgery Postoperative (Visit 6) 3-4 months after surgery

Postoperatively, logMAR visual acuity will be recorded at every visit and non-cycloplegic refraction will be carried out at Visit 5 and Visit 6.

ELIGIBILITY:
Inclusion Criteria:

1. Eyes with significant cataract and suitable for phacoemulsification and primary implantation of posterior chamber intraocular lens.
2. Cataract as the only ophthalmic pathology causing significant visual impairment.
3. Axial length less than 22mm or more than 25mm, as measured by Zeiss IOL Master.
4. Evidence of a personally signed and dated informed consent document indicating the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
5. Patient is willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

1. Presence of other ophthalmic pathology causing visual impairment: amblyopia, glaucoma, optic neuropathy, age related macular degeneration, macular oedema, retinal detachment, proliferative diabetic retinopathy, ocular inflammation.
2. Previous intraocular or corneal surgery (including refractive surgery).
3. Corneal opacities or irregularities: previous scarring, dystrophy, ectasia
4. Corneal astigmatism greater than 1.5 dioptres.
5. Axial length unable to be measured by the Zeiss IOL master.
6. Other ocular surgery at time of cataract extraction.
7. Uncontrolled diabetes.
8. Any neurological condition which may interfere with performance of required tests.
9. Other severe acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.

Surgical exclusion criteria

The patient will not be included in the study if any of the following complications are encountered during surgery:

1. Inability to achieve secure 'in-the-bag' placement of the IOL (i.e. due to posterior capsule rupture, radial tear in capsulorhexis, vitreous loss, zonular rupture)
2. Use of corneal sutures.
3. Multiple operative procedures at the time of IOL implantation.

   Post-implantation exclusion criteria:
4. Haptic not in the capsular bag.
5. Decentration of the IOL of more than 1.0mm.
6. Other ocular pathology causing visual impairment that were not apparent prior to surgery (e.g. age related macular degeneration, macular oedema, glaucoma, retinal detachment).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2005-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mean absolute error (MAE) which is calculated by subtracting the intended formula-derived preoperative refractive error from the actual postoperative refractive error.

CONTACTS AND LOCATIONS:
Overall Officials: Zainah Alsagoff, FRCSEd, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore